CLINICAL TRIAL: NCT04736888
Title: Comparison of Extended Reality and Conventional Methods of Basic Life Support Training: Protocol for a Multinational Pragmatic Clinical Trial (XR BLS Trial)
Brief Title: Effectiveness of Extended Reality CPR Training Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Children's Hospital Los Angeles (Other); Royal Manchester Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Dong Keon Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CBS2.0
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Basic Cardiac Life Support; Virtual Reality
Keywords: Cardiopulmonary resuscitation; Basic Cardiac Life Support; Virtual Reality; Extended Reality; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional group (Sham Comparator): Conventional CPR training consists of a BLS video and a manikin equipped with a feedback device.
  Interventions: Other: conventional CPR training
- XR group (Active Comparator): The XR group participants will be provided training via the XR BLS module and are allotted an additional 2 minutes that is needed to adapt to the XR equipment.
  Interventions: Other: extended-reality CPR training

INTERVENTIONS:
Other: extended-reality CPR training — extended-reality technologies based CPR training module
  Arms: XR group
Other: conventional CPR training — conventional CPR training with video
  Arms: Conventional group

SUMMARY:
The aim of this study is to explore the efficacy and safety of the extended reality (XR)-based basic life support (BLS) training.

DETAILED DESCRIPTION:
Conventional CPR training is based on the use of a manikin and a training video. Though several feedback devices have been developed to improve the effectiveness of the training, they were neither realistic nor immersive. In addition, in conventional training programs, trainees are constrained in terms of time and location, as they are usually kept to a schedule.

Virtual reality (VR) technology, which was designed to maximize immersion, could be used to overcome those limitations, which in turn may improve the effectiveness of CPR training. However, even with VR technology, procedures such as chest compressions, ventilation, and defibrillation cannot be implemented as in the real world. Extended reality (XR), which combines the virtual and real worlds, could overcome these limitations by facilitating the use of real-world manikins in the virtual environment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are not healthcare providers and are 18 years old or older

Exclusion Criteria:

Participants who

* are not capable of performing either the training or the CPR test due to physical or cognitive limitations
* have upper extremity injuries
* are pregnant
* experience dizziness, headache, or motion sickness during the 2-minute XR device adaptation period that prevents them from participating in the simulation study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
mean compression depth, mm | Test sessions on day 1 (during 5 minutes) after 1 hour training
  compression depth

SECONDARY OUTCOMES:
the total number of chest compressions (n) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  The total number of chest compressions
the mean chest compression depth(mm) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  compression depth between 5cm and 6cm
correct hand position (n, percent) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  The American Heart Association (AHA) guidelines describe the correct hand position for chest compression as the lower half of the victim's sternum in the centre of the chest, between the nipples.
adequate compression depth (n, percent) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  compression depth between 5cm and 6cm
compression and full release (n, percent) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  full release after chest compression
mean compression rate (number per minute) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  mean compression rate
adequate compression rate (percent) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  compression rate between 100 and 120 per minute
adequate compression depth and rate (percent) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  adequate compression death and rate, simultaneously
hands-off time (sec) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  Interruptions of chest compressions during cardiopulmonary resuscitation
The time interval from arrival on the scene to the first chest compression (sec) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  The time interval from arrival on the scene to the first chest compression.
AED use | Test sessions on day 1 (during 5 minutes) after 1 hour training
  Done/Not done
Correct AED use | Test sessions on day 1 (during 5 minutes) after 1 hour training
  Yes/No
Time from powering on the AED to defibrillation (sec) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  Time from powering on the AED to defibrillation (sec)
Time from checking for a response to defibrillation (sec) | Test sessions on day 1 (during 5 minutes) after 1 hour training
  Time from checking for a response to defibrillation (sec)

CONTACTS AND LOCATIONS:
Overall Officials: You Hwan Jo, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semeraro F, Frisoli A, Loconsole C, Banno F, Tammaro G, Imbriaco G, Marchetti L, Cerchiari EL. Motion detection technology as a tool for cardiopulmonary resuscitation (CPR) quality training: a randomised crossover mannequin pilot study. Resuscitation. 2013 Apr;84(4):501-7. doi: 10.1016/j.resuscitation.2012.12.006. Epub 2012 Dec 10. PMID 23238423
- [Background] Semeraro F, Taggi F, Tammaro G, Imbriaco G, Marchetti L, Cerchiari EL. iCPR: a new application of high-quality cardiopulmonary resuscitation training. Resuscitation. 2011 Apr;82(4):436-41. doi: 10.1016/j.resuscitation.2010.11.023. Epub 2011 Jan 11. PMID 21227560
- [Background] Semeraro F, Frisoli A, Bergamasco M, Cerchiari EL. Virtual reality enhanced mannequin (VREM) that is well received by resuscitation experts. Resuscitation. 2009 Apr;80(4):489-92. doi: 10.1016/j.resuscitation.2008.12.016. Epub 2009 Feb 8. PMID 19203823
- [Background] Iwashyna TJ. Survivorship will be the defining challenge of critical care in the 21st century. Ann Intern Med. 2010 Aug 3;153(3):204-5. doi: 10.7326/0003-4819-153-3-201008030-00013. No abstract available. PMID 20679565
- [Background] Grasner JT, Lefering R, Koster RW, Masterson S, Bottiger BW, Herlitz J, Wnent J, Tjelmeland IB, Ortiz FR, Maurer H, Baubin M, Mols P, Hadzibegovic I, Ioannides M, Skulec R, Wissenberg M, Salo A, Hubert H, Nikolaou NI, Loczi G, Svavarsdottir H, Semeraro F, Wright PJ, Clarens C, Pijls R, Cebula G, Correia VG, Cimpoesu D, Raffay V, Trenkler S, Markota A, Stromsoe A, Burkart R, Perkins GD, Bossaert LL; EuReCa ONE Collaborators. EuReCa ONE-27 Nations, ONE Europe, ONE Registry: A prospective one month analysis of out-of-hospital cardiac arrest outcomes in 27 countries in Europe. Resuscitation. 2016 Aug;105:188-95. doi: 10.1016/j.resuscitation.2016.06.004. Epub 2016 Jun 16. PMID 27321577
- [Background] Deakin CD. The chain of survival: Not all links are equal. Resuscitation. 2018 May;126:80-82. doi: 10.1016/j.resuscitation.2018.02.012. Epub 2018 Feb 19. PMID 29471008
- [Background] Brady WJ, Mattu A, Slovis CM. Lay Responder Care for an Adult with Out-of-Hospital Cardiac Arrest. N Engl J Med. 2019 Dec 5;381(23):2242-2251. doi: 10.1056/NEJMra1802529. No abstract available. PMID 31800989
- [Background] Ro YS, Shin SD, Song KJ, Hong SO, Kim YT, Cho SI. Bystander cardiopulmonary resuscitation training experience and self-efficacy of age and gender group: a nationwide community survey. Am J Emerg Med. 2016 Aug;34(8):1331-7. doi: 10.1016/j.ajem.2015.12.001. Epub 2015 Dec 7. PMID 27037129
- [Background] Andrews C, Southworth MK, Silva JNA, Silva JR. Extended Reality in Medical Practice. Curr Treat Options Cardiovasc Med. 2019 Mar 30;21(4):18. doi: 10.1007/s11936-019-0722-7. PMID 30929093
- [Background] Nas J, Thannhauser J, Vart P, van Geuns RJ, Muijsers HEC, Mol JQ, Aarts GWA, Konijnenberg LSF, Gommans DHF, Ahoud-Schoenmakers SGAM, Vos JL, van Royen N, Bonnes JL, Brouwer MA. Effect of Face-to-Face vs Virtual Reality Training on Cardiopulmonary Resuscitation Quality: A Randomized Clinical Trial. JAMA Cardiol. 2020 Mar 1;5(3):328-335. doi: 10.1001/jamacardio.2019.4992. PMID 31734702
- [Background] Anderson R, Sebaldt A, Lin Y, Cheng A. Optimal training frequency for acquisition and retention of high-quality CPR skills: A randomized trial. Resuscitation. 2019 Feb;135:153-161. doi: 10.1016/j.resuscitation.2018.10.033. Epub 2018 Nov 2. PMID 30391370
- [Background] Bylow H, Karlsson T, Claesson A, Lepp M, Lindqvist J, Herlitz J. Self-learning training versus instructor-led training for basic life support: A cluster randomised trial. Resuscitation. 2019 Jun;139:122-132. doi: 10.1016/j.resuscitation.2019.03.026. Epub 2019 Mar 26. PMID 30926451
- [Background] Roppolo LP, Pepe PE, Campbell L, Ohman K, Kulkarni H, Miller R, Idris A, Bean L, Bettes TN, Idris AH. Prospective, randomized trial of the effectiveness and retention of 30-min layperson training for cardiopulmonary resuscitation and automated external defibrillators: The American Airlines Study. Resuscitation. 2007 Aug;74(2):276-85. doi: 10.1016/j.resuscitation.2006.12.017. Epub 2007 Apr 23. PMID 17452070
- [Background] Zapletal B, Greif R, Stumpf D, Nierscher FJ, Frantal S, Haugk M, Ruetzler K, Schlimp C, Fischer H. Comparing three CPR feedback devices and standard BLS in a single rescuer scenario: a randomised simulation study. Resuscitation. 2014 Apr;85(4):560-6. doi: 10.1016/j.resuscitation.2013.10.028. Epub 2013 Nov 8. PMID 24215730
- [Background] Park S, Lee G. Full-immersion virtual reality: Adverse effects related to static balance. Neurosci Lett. 2020 Aug 10;733:134974. doi: 10.1016/j.neulet.2020.134974. Epub 2020 Apr 12. PMID 32294492
- [Background] Edelson DP, Sasson C, Chan PS, Atkins DL, Aziz K, Becker LB, Berg RA, Bradley SM, Brooks SC, Cheng A, Escobedo M, Flores GE, Girotra S, Hsu A, Kamath-Rayne BD, Lee HC, Lehotsky RE, Mancini ME, Merchant RM, Nadkarni VM, Panchal AR, Peberdy MAR, Raymond TT, Walsh B, Wang DS, Zelop CM, Topjian AA; American Heart Association ECC Interim COVID Guidance Authors. Interim Guidance for Basic and Advanced Life Support in Adults, Children, and Neonates With Suspected or Confirmed COVID-19: From the Emergency Cardiovascular Care Committee and Get With The Guidelines-Resuscitation Adult and Pediatric Task Forces of the American Heart Association. Circulation. 2020 Jun 23;141(25):e933-e943. doi: 10.1161/CIRCULATIONAHA.120.047463. Epub 2020 Apr 9. No abstract available. PMID 32270695
- [Background] Nolan JP, Monsieurs KG, Bossaert L, Bottiger BW, Greif R, Lott C, Madar J, Olasveengen TM, Roehr CC, Semeraro F, Soar J, Van de Voorde P, Zideman DA, Perkins GD; European Resuscitation Council COVID-Guideline Writing Groups. European Resuscitation Council COVID-19 guidelines executive summary. Resuscitation. 2020 Aug;153:45-55. doi: 10.1016/j.resuscitation.2020.06.001. Epub 2020 Jun 7. PMID 32525022
- [Background] Craig-Brangan KJ, Day MP. Update: AHA guidelines for CPR and emergency cardiovascular care. Nursing. 2020 Jun;50(6):58-61. doi: 10.1097/01.NURSE.0000659320.66070.a9. PMID 32453156
- [Background] Riggs M, Franklin R, Saylany L. Associations between cardiopulmonary resuscitation (CPR) knowledge, self-efficacy, training history and willingness to perform CPR and CPR psychomotor skills: A systematic review. Resuscitation. 2019 May;138:259-272. doi: 10.1016/j.resuscitation.2019.03.019. Epub 2019 Mar 27. PMID 30928504
- [Background] Stiell IG, Brown SP, Nichol G, Cheskes S, Vaillancourt C, Callaway CW, Morrison LJ, Christenson J, Aufderheide TP, Davis DP, Free C, Hostler D, Stouffer JA, Idris AH; Resuscitation Outcomes Consortium Investigators. What is the optimal chest compression depth during out-of-hospital cardiac arrest resuscitation of adult patients? Circulation. 2014 Nov 25;130(22):1962-70. doi: 10.1161/CIRCULATIONAHA.114.008671. Epub 2014 Sep 24. PMID 25252721
- [Derived] Lee DK, Im CW, Jo YH, Chang T, Song JL, Luu C, Mackinnon R, Pillai S, Lee CN, Jheon S, Ahn S, Won SH. Comparison of extended reality and conventional methods of basic life support training: protocol for a multinational, pragmatic, noninferiority, randomised clinical trial (XR BLS trial). Trials. 2021 Dec 20;22(1):946. doi: 10.1186/s13063-021-05908-z. PMID 34930418